CLINICAL TRIAL: NCT05893719
Title: First Prospective, Single-arm, Multicentre Study to Evaluate the Safety and Efficacy of the Overall Thrombectomy System for Stroke: iNedit, iNdeep and iNtercept in Patients With Acute Ischemic Stroke.
Brief Title: Prospective, Multicentre Study to Evaluate the Thrombectomy System for Stroke: iNedit, iNdeep and iNtercept
Acronym: SEMTiC
Status: Completed | Type: Observational
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: SEMTiC-01
Record Dates: First submitted 2022-07-21; First posted 2023-06-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Mechanical Neurothrombectomy; Ischemia
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: iNedit, iNdeep, iNtercept: Study devices
  Interventions: Device: iNedit, iNdeep, iNtercept

INTERVENTIONS:
Device: iNedit, iNdeep, iNtercept — Patients to undergo mechanical thrombectomy with iNedit, iNdeep and iNtercept

SUMMARY:
First prospective, single-arm, multicentre study to evaluate the safety and efficacy of the overall stroke thrombectomy system: iNedit, iNdeep and iNtercept in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
This is a prospective, multicentre, single-arm and open-label clinical safety and efficacy research.

The purpose of the study is to evaluate the safety and efficacy of the three devices designed by iVascular for neurothrombectomy (iNedit, iNdeep and iNtercept) used together as a tool to facilitate the placement of the stent retriever and apply temporary restriction of blood flow in patients who have suffered a stroke and who undergo mechanical thrombectomy due to acute large vessel occlusion (LVO), presented within 8 hours from symptoms onset (the last time the patient was seen well).

Being a mechanical thrombectomy the procedure by which the thrombus that occludes a cerebral vessel is accessed. It is accessed through an endovascular catheter, inserted through the femoral artery, for disruption or removal.

ELIGIBILITY:
Inclusion Criteria:

Clinical:

1. Age ≥18
2. Informed consent signed by the patient or their representative; to use the patient's data
3. Focal disabling neurologic deficit consistent with acute cerebral ischemia.
4. Baseline NIHSS obtained before procedure of ≥6 points and ≤25 points.
5. Pre-stroke mRS score ≤2.
6. Planning to start treatment within 24 hours of symptoms onset, defined as the last time when the patient was seen well (the start of the procedure is defined as arterial puncture).

Neuroimaging criteria:

1. Occlusion (TICI 0 or TICI 1) of the internal intracranial carotid artery, M1 and M2 segments of the middle cerebral artery and T carotid artery, suitable for mechanical thrombectomy confirmed by conventional angiography.
2. For patients treated ≤8 hours:

   a) Score 6 to 10 on ASPECTS scale (Alberta Stroke Program Early CT Score).

   For patients treated between 8 and 24 hours:

   a) "Target Mismatch Profile" on CT perfusion or MRI (ischemic core volume is <70mL, mismatch ratio is >1,8 and mismatch volume is >15 mL).
3. Ability to obtain selective angiography by catheterisation of the target artery.

Exclusion Criteria:

Clinical:

1. Patient has suffered a stroke in the past one year.
2. Occlusion (TICI 0 or TICI 1) in vertebrobasilar territory.
3. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
4. Known hemorrhagic diathesis, coagulaion factor deficiency or oral anti-vitamin K anticoagulant therapy with an INR >3.0.
5. Blood glucose <50 mg/dl or >400 mg/dl. NOTE: If blood glucose can be successfully reduced and maintained at an acceptable level by administering the medication recommended by the ESO (European Stroke Organisation) in its guidelines, the patient may be included.
6. Severe sustained hypertension (systolic pressure >185 mm Hg or diastolic pressure >110 mm Hg). NOTE: If blood pressure can be successfully reduced and maintained at an acceptable level by administering the medication recommended by the ESO (European Stroke Organisation) in its guidelines (also IV infusion of antihypertensives), the patient may be included.
7. Serious advanced or terminal illness with anticipated life expectancy of less than six months.
8. History of life-threatening allergy (more than rash) to contrast medium.
9. Known allergy to nickel, prior to treatment.
10. Known renal insufficiency with creatinine ≥3 mg/dl or Glomerular Filtration Rate (GFR) <30 mL/min.
11. Cerebral vasculitis.
12. Known current cocaine use.
13. Patient who is participating, at the time of inclusion, in a study with a device or drug that could affect this study.
14. Patients who are unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitors from overseas).

Neuroimaging criteria:

1. CT or MRI evidence of hemorrhage (the presence of microbleeds is allowed).
2. Significant mass effect with midline shift.
3. Evidence of complete occlusion, high-grade stenosis or arterial dissection in the extracranial or petrous segment of the internal carotid artery (TANDEM lesions).
4. Patients with known or suspected underlying intracranial atherosclerotic lesions responsible for the target occlusion.
5. Patients with occlusions in multiple vascular territories (e.g. bilateral anterior circulation or anterior/posterior circulation).
6. Evidence of intracranial tumour with the exception of asymptomatic meningiomas with no mass effect.
7. Presumed septic embolism with suspected aortic dissection or suspicion of bacterial endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present acute stroke, attributable to occlusion of the internal carotid artery, M1 or M2 segments of the middle cerebral artery, and who are not suitable to receive IV rtPA or who have already received IV rtPA treatment without sufficient recanalization, within 24 hours from symptoms onset (or the last time they were seen well) to groin puncture in the catheterisation laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Performance Success | In the course of endovascular procedure, evaluated immediately after it.
  To assess the ability of the system to successfully perform a neurothrombectomy using the three devices to be evaluated and with ≤3 insertions (passes) of the stent retriever.
MAE | 24 hours (-8/+12 hours)
  All serious adverse events following the intervention or until an alternative stroke treatment is started, whichever occurs first.
Mortality | 90 days
  All-cause mortality

SECONDARY OUTCOMES:
Clinical progress | 90 days
  Good functional clinical progress (modified Rankin scale 0-2)
Proportion of patients with rapid neurological improvement | 24 hours after treatment
  Proportion of patients with rapid neurological improvement (more than 4 points on the NIHSS scale, or NIHSS ≤4)
Reduction of NIHSS scale | At 72 hours or at the time of discharge, whichever occurs first.
  Proportion of patients with a reduction of ≥8 points on the NIHSS scale or NIHSS 0-1
Procedure duration | In the course of endovascular procedure, evaluated immediately after it.
  Procedure duration defined as the time from puncture to when grade ≥2b is reached on the mTICI scale with less than three passes or, if not achieved, until the final angiogram.
Number of passes with the device until recanalization. | In the course of endovascular procedure, evaluated immediately after it.
  Number of passes with the device until recanalization.
Percentage of effective recanalization in a first pass. | In the course of endovascular procedure, evaluated immediately after it.
  Percentage of effective recanalization in a first pass.
Rate of cases that reached the occlusion and allowed the performance of the trombectomy. | In the course of endovascular procedure, evaluated immediately after it.
  Rate of cases where the microcatheter and the distal access balloon catheter reached the occlusion in the main vessel to allow navigation and deployment of the stent retriever to carry out the neurothrombectomy.
Assessment of intracranial haemorrhage (ICH) | 24 (-8/+12) hours
  Assessment of intracranial haemorrhage (ICH); any symptomatic or asymptomatic intracranial haemorrhage assessed by magnetic resonance imaging (MRI) /computed tomography (CT).
Neurological deterioration | 24 (-8/+12) hours.
  Classification of neurological deterioration of ≥4 points on the NIHSS scale
Embolization rate | In the course of endovascular procedure, evaluated immediately after it.
  Embolization rate in a previously non-involved territory on cerebral angiography.
Mortality rate | 3 days (+/-24) hours
  Mortality rate related to the procedure
Procedure complication rate | In the course of endovascular procedure, evaluated immediately after it.
  Procedure complication rate: arterial perforation, arterial dissection and vasospasm in the target vessel and embolization in a previously non-involved vascular territory.
Rate of infarction in a previously non-involved vascular territory | 24 hours.
  Rate of infarction in a previously non-involved vascular territory, as evaluated by imaging (MRI/CT).

CONTACTS AND LOCATIONS:
Locations (18):
- Hospital AZ Groeninge, Kortrijk, Belgium
- Germany (3):
  - Hospital Klinikum Ludwigsburg, Ludwigsburg
  - Hospital LMU Klinikum, Munich
  - Hospital Klinikum Nürnberg, Nuremberg
- Spain (14):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital de Cruces, Barakaldo
  - Hospital de la Vall d'Hebrón, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital GermansTrias i Pujol, Barcelona
  - Hospital Reina Sofia de Córdoba, Córdoba
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico de Valencia, Valencia
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] San Roman L, Gramegna LL, Pich S, Domingo-Rodriguez L, Duran M, Duocastella L, Macho J. First prospective, single-arm, multicenter study to evaluate safety and efficacy of the overall thrombectomy system -iNedit, iNdeep, and iNtercept- for acute ischemic stroke. Rationale beyond the study. Front Neurol. 2025 Mar 5;16:1537008. doi: 10.3389/fneur.2025.1537008. eCollection 2025. PMID 40134692
- [Result] Tomasello A, Gramegna LL, Vega P, Castano C, Moreu M, Dominguez C, Macho J. Mechanical thrombectomy with a new intermediate balloon catheter combining the BGC and DAC features: Initial clinical experience with the iNedit device. Interv Neuroradiol. 2023 Oct 17:15910199231207407. doi: 10.1177/15910199231207407. Online ahead of print. PMID 37847747